CLINICAL TRIAL: NCT00441467
Title: An Open-Label Phase 2 Study of the Efficacy and Safety of Glufosfamide in Previously Treated Advanced Soft Tissue Sarcoma
Brief Title: Safety and Efficacy Study of Glufosfamide in Previously Treated Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eleison Pharmaceuticals LLC. (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-305
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — beta-D-glucosylisophosphoramide mustard

ARMS (1):
- Glufosfamide (Experimental): Glufosfamide
  Interventions: Drug: Glufosfamide

INTERVENTIONS:
Drug: Glufosfamide — 5000 mg/m2 of glufosfamide on Day 1 of each three-week cycle for up to 6 cycles.

SUMMARY:
Primary Objective:

1. To evaluate the efficacy of glufosfamide in subjects with advanced soft tissue sarcoma as measured by objective response rate

Secondary Objectives:

1. To evaluate the efficacy of glufosfamide in subjects with advanced soft tissue sarcoma as measured by duration of response, progression-free survival and overall survival
2. To evaluate the safety of glufosfamide in subjects with advanced soft tissue sarcoma

Exploratory Objectives:

1. To evaluate the biological effect of glufosfamide on the metabolic profile in subjects with advanced soft tissue sarcomas, as determined by FDG-PET
2. To correlate efficacy endpoints with expression of tumor-associated glucose transporter proteins

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Pathologically confirmed diagnosis of soft tissue sarcoma
* Locally advanced unresectable or metastatic disease with no standard curative therapy available that has progressed since the most recent therapy
* Measurable disease by RECIST criteria with at least one target lesion
* 1 or 2 prior chemotherapy/systemic therapy regimens for advanced disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2
* A minimum of 3 weeks between prior chemotherapy, radiation therapy, immunotherapy, or other anti-tumor therapy and study entry
* Recovered from reversible toxicities of prior therapy
* Hemoglobin ≥ 9.0 g/dL, neutrophils ≥ 1,500/µL, platelets ≥ 100,000/µL
* Total bilirubin ≤ 1.5-fold ULN, AST/ALT ≤ 2.5-fold ULN (≤ 5-fold if liver metastases)
* Normal creatinine clearance (≥85 mL/min for men and ≥75 mL/min for women; calculated by Cockcroft-Gault formula
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) from entry into the study through 6 months after the last dose

Exclusion Criteria:

* Soft tissue sarcoma of the following subtypes: gastrointestinal stromal tumor (GIST), alveolar soft parts sarcoma, hemangiopericytoma and Kaposi's sarcoma
* Most recent relapse occurring during treatment with ifosfamide within 4 weeks of last dose
* Symptomatic brain or leptomeningeal metastases
* Active clinically significant infection requiring antibiotics
* Recent (one year) history or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4), particularly coronary artery disease, arrhythmias or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, cerebrovascular accident or congestive heart failure
* Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years
* Major surgery within 3 weeks of the start of study treatment, without complete recovery
* Females who are pregnant or breast-feeding
* Participation in an investigational drug or device study within 21 days of study entry
* Concomitant disease or condition that could interfere with the conduct of the study, or that in the opinion of the investigator would pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, PhD, Principal Investigator — University of Arizona; David Mendelson, MD, Principal Investigator — Premiere Oncology of Arizona; Douglas Adkins, MD, Principal Investigator — Washington University School of Medicine, Division of Oncology; Gina D'Amato, MD, Principal Investigator — H. Lee Moffitt Cancer Center; Gerald Rosen, MD, Principal Investigator — St. Vincent's Comprehensive Cancer Center; Claire Verschraegen, MD, Principal Investigator — University of New Mexico Cancer Center; Kristen Ganjoo, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Stanford Cancer Center, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, Division of Oncology, St Louis, Missouri
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - St. Vincent's Comprehensive Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glufosfamide
Started | 22
2 Cycles | 17
4 Cycles | 7
Completed | 4
Not Completed | 18
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 3
Not completed — Progressive disease | 9

BASELINE CHARACTERISTICS:
Arm/Group | Glufosfamide
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 53.5 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The event rate was the response rate (complete and partial response) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.0). The associated 95% exact binomial confidence intervals were calculated.
Time Frame: Tumor assessments were performed at baseline and every 6 weeks until disease progression was documented.
Population: Patients receiving glufosfamide with a post treatment imaging assessment
Measure: Number; unit: participants
Arm/Group | Glufosfamide
Number analyzed (Participants) | 19
participants
  Partial response | 1
  Stable disease | 7
  Progressive disease | 11

2. Secondary Outcome: Progression-free Survival
Time Frame: All subjects were followed regularly until glufosfamide discontinuation, tumor progression or additional antitumor therapy was started and then were followed for survival at 3 month intervals for the first year and once every year thereafter until death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glufosfamide
Number analyzed (Participants) | 22
months | 1.3 [1.3 to 3.9]

3. Secondary Outcome: Overall Survival
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glufosfamide
Number analyzed (Participants) | 22
months | 10.5 [6.3 to 13.6]

ADVERSE EVENTS:
Arm/Group | Glufosfamide
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glufosfamide (N=22)
Renal failure (Renal and urinary disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Intractable nausea and vomiting (Gastrointestinal disorders) | 1 (2)
Sarcoma site hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glufosfamide (N=22)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anemia aggravated (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Depression aggravated (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal bloating (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Constipation agravated (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (20)
Nausea aggravated (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain aggravated (Musculoskeletal and connective tissue disorders) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 5 (6)
Fatigue aggravated (General disorders) | 3 (3)
General body pain (General disorders) | 2 (2)
Weakness (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No